CLINICAL TRIAL: NCT03231345
Title: Ultrasound-guided Placement of Peripheral Intravenous Lines in the Internal Jugular Vein.
Brief Title: Ultrasound-guided Peripheral IJ Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center of Southern Nevada (Other)
Responsible Party: Principal Investigator, Joseph (Tony) Zitek, MD, MD, Assistant Research Director, Emergency Medicine Residency Program, University Medical Center of Southern Nevada
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 16.08.002
Record Dates: First submitted 2017-07-22; First posted 2017-07-27 (Actual); Results first posted 2019-01-15 (Actual); Last update posted 2019-01-15 (Actual); Status verified 2019-01

CONDITIONS: IV Access
Keywords: Peripheral IV; Internal jugular vein; IJ; Peripheral IJ; Ultrasound-guided IJ
MeSH Terms: interventions — Ultrasonography

STUDY DESIGN:
Intervention Model Description: This study utilizes a convenience sample of patient who have difficult venous access with at least 2 attempts by nursing to achieve venous access. The patient will be consented and a physician placed ultrasound-guided peripheral IV will be placed in the internal jugular vein.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- US guided IJ (Experimental): A physician placed ultrasound-guided IV in the internal jugular vein
  Interventions: Procedure: US guided IJ; Device: Ultrasound

INTERVENTIONS:
Procedure: US guided IJ — IV catheter placement
  Other Names: Ultrasound-guided Internal Jugular vein
Device: Ultrasound — Ultrasound-guided Internal Jugular vein

SUMMARY:
Difficult venous access in some patients such as those with obesity, IV drug use, chronic illness, or vascular pathology often causes increased discomfort and delayed patient care due to multiple attempts to gain venous access. If access is achieved at all, it usually results in a much smaller catheter than needed to provide optimal care for the patient. Ultrasound-guided placement of a peripheral IV in the internal jugular vein is common in the investigators' emergency department and is gaining popularity across the US. This study investigates the utility and safety of placing an ultrasound-guided peripheral IV catheter in the internal jugular vein.

DETAILED DESCRIPTION:
Intravenous access in the emergency department (ED) patient is essential for medication delivery, IV fluid resuscitation, rapid serum laboratory diagnostics, and administration of IV contrast for CT scans. Some patients, such as those with obesity, IV drug abuse, chronic illnesses, or vascular pathology may have difficult IV access. These patients are problematic for the busy ED nurse and physician as this can lead to a time consuming process, which slows efficiency and patient care.

Previously, patients with difficult IV access often required central venous catheterization, a procedure that can result in a number of serious complications (1). More recently, ultrasound guidance has been touted as an effective means to achieve peripheral IV access on these patients (2). In one study (2), there was a 73% first attempt cannulation rate, which seems respectable, but not excellent. Additionally, 8% of the successful IVs failed within one hour (2). Another study compared ultrasonographically guided peripheral IVs to non-ultrasonographically guided IVs, and it found that using ultrasound did not decrease the amount of time or the number of attempts it took to successfully place a peripheral IV (3). Although ultrasound-guided peripheral IV's have a role, there remains room for improvement in being able to achieve rapid IV access in those patients who need IV access on an urgent basis.

It seems that we still have room to improve our ability to obtain difficult IV access, and a relatively new technique may be the answer. Ultrasound guided IVs are typically attempted in the upper extremities, targeting the brachial or basilic veins, but a recently described technique --- the "peripheral IJ" --- involves placement of a peripheral IV catheter in the internal jugular vein (4,5).

The peripheral IJ is gaining popularity in the investigators' ED as a solution to the difficult vascular access patient. In the investigators' clinical experience, it is a quick and easy procedure that is also safe, tolerated well by patients, and requires few resources. Several small studies have concluded that this is a fast and safe procedure and a feasible alternative to central access in the difficult vascular access patient (4-7). These studies mention the theoretical risks as being similar to central venous access such as carotid artery puncture, hematoma, pneumothorax, and line infection, however none of these have actually been reported (4-7). Therefore, we seek primarily to determine the average number of attempts to cannulation for ultrasound-guided peripheral IJ placement. Secondarily, we wish to determine: 1) the prevalence of potential complications related to this procedure 2) the average time it takes the emergency physician to complete the procedure 3) the patient's satisfaction with the procedure. We will compare the data from this study to the published data for other types of ultrasound-guided peripheral IVs.

ELIGIBILITY:
Inclusion Criteria:

* At least 2 unsuccessful attempts at peripheral IV access by ED nursing
* Age 18 or older

Exclusion Criteria:

* Critically ill patients with clinical indications for emergent central venous access.
* Overlying skin infection
* External jugular vein easily visible for cannulation
* Patient in law enforcement custody
* Patient who is known to be pregnant or self identifies as pregnant
* Patient lacking decision making capacity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2016-08-18 (Actual); Primary Completion 2017-09-06 (Actual); Study Completion 2018-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph A Zitek, MD, Principal Investigator — UMCSN
Locations (1):
- University Medical Center of Southen Nevada, Las Vegas, Nevada, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kornbau C, Lee KC, Hughes GD, Firstenberg MS. Central line complications. Int J Crit Illn Inj Sci. 2015 Jul-Sep;5(3):170-8. doi: 10.4103/2229-5151.164940. PMID 26557487
- [Background] Keyes LE, Frazee BW, Snoey ER, Simon BC, Christy D. Ultrasound-guided brachial and basilic vein cannulation in emergency department patients with difficult intravenous access. Ann Emerg Med. 1999 Dec;34(6):711-4. doi: 10.1016/s0196-0644(99)70095-8. PMID 10577399
- [Background] Stein J, George B, River G, Hebig A, McDermott D. Ultrasonographically guided peripheral intravenous cannulation in emergency department patients with difficult intravenous access: a randomized trial. Ann Emerg Med. 2009 Jul;54(1):33-40. doi: 10.1016/j.annemergmed.2008.07.048. Epub 2008 Sep 27. PMID 18824276
- [Background] Teismann NA, Knight RS, Rehrer M, Shah S, Nagdev A, Stone M. The ultrasound-guided "peripheral IJ": internal jugular vein catheterization using a standard intravenous catheter. J Emerg Med. 2013 Jan;44(1):150-4. doi: 10.1016/j.jemermed.2012.02.044. Epub 2012 May 11. PMID 22579025
- [Background] Butterfield M, Abdelghani R, Mohamad M, Limsuwat C, Kheir F. Using Ultrasound-Guided Peripheral Catheterization of the Internal Jugular Vein in Patients With Difficult Peripheral Access. Am J Ther. 2017 Nov/Dec;24(6):e667-e669. doi: 10.1097/MJT.0000000000000357. PMID 26469683
- [Background] Kiefer D, Keller SM, Weekes A. Prospective evaluation of ultrasound-guided short catheter placement in internal jugular veins of difficult venous access patients. Am J Emerg Med. 2016 Mar;34(3):578-81. doi: 10.1016/j.ajem.2015.11.069. Epub 2015 Dec 4. PMID 26776533
- [Background] Zwank MD. Ultrasound-guided catheter-over-needle internal jugular vein catheterization. Am J Emerg Med. 2012 Feb;30(2):372-3. doi: 10.1016/j.ajem.2011.08.013. Epub 2011 Oct 26. No abstract available. PMID 22033389
- [Background] Ash AJ, Raio C. Seldinger Technique for Placement of "Peripheral" Internal Jugular Line: Novel Approach for Emergent Vascular Access. West J Emerg Med. 2016 Jan;17(1):81-3. doi: 10.5811/westjem.2015.11.28726. Epub 2016 Jan 12. PMID 26823937

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | US Guided IJ
Started | 35
Completed | 35
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | US Guided IJ
Number analyzed (Participants) | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.2 (15.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 10
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 14
  African American | 14
  Hispanic | 6
  Asian | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 35

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Successful Cannulation of the Internal Jugular Vein
Description: The primary study endpoint is successful cannulation vs failure to cannulate the internal jugular vein.
Time Frame: Less than 20 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | US Guided IJ
Number analyzed (Participants) | 35
Participants | 34

2. Secondary Outcome: Prevalence of Complications Related to Cannulation of the Internal Jugular Vein.
Description: Percentage of Participants with successfully placed lines with a complication
Time Frame: 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | US Guided IJ
Number analyzed (Participants) | 34
Participants | 1

3. Secondary Outcome: The Median Time Required for Cannulation of the Internal Jugular Vein by an Emergency Physician.
Description: The median time it took an Emergency Physician from needle puncture to cannulation in minutes
Time Frame: Less than 20 minutes
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | US Guided IJ
Number analyzed (Participants) | 34
minutes | 3.1 [0.98 to 4.2]

ADVERSE EVENTS:
Time Frame: We monitored for adverse events throughout the patient's hospitalization, the length of which ranged from a few hours to a maximum of 2 weeks.
Description: The adverse events that we tracked included local hematoma, pneumothorax, arterial puncture, bacteremia/line infection, and line thrombus. Trained research assistants watched line placement to assess for these complications. They also rechecked the line 1 hour after placement, and then once every 24 hours until the line was removed. They also checked the results of CXRs to look for pneumothoraces, and they checked blood cultures results.
Arm/Group | US Guided IJ
All-Cause Mortality (participants affected / at risk) | 0/35
Serious Adverse Events (participants affected / at risk) | 0/35
Other Adverse Events (participants affected / at risk) | 1/35
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | US Guided IJ (N=35)
Complications from IV line placement (Vascular disorders) | 1 (1) — The only complication found was a local hematoma.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2017-04-01): https://cdn.clinicaltrials.gov/large-docs/45/NCT03231345/Prot_000.pdf